CLINICAL TRIAL: NCT03993652
Title: Kids FIRST: Development and Feasibility of a Family-based Intervention to Reduce Snacking and Screen Time in Children
Brief Title: Kids FIRST: Family-based Intervention to Reduce Snacking and Screen Time in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Natalie Pearson, Senior Research Associate in Physical Activity and Public Health, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PG/12/70/29777
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Sedentary Lifestyle; Sedentary Behavior; Diet Habit
MeSH Terms: conditions — Sedentary Behavior; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: 4-arm intervention. 3 interventions that received the same model but tailored to behavioural target. control group received no treatment
Who Masked: Investigator
Masking Description: schools were blinded to study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Screen-time and Snacking (Experimental): Aim: to reduce both screen-time and unhealthy snacking
  Interventions: Behavioral: Kids FIRST
- Screen-time only (Experimental): Aim: to reduce screen-time only
  Interventions: Behavioral: Kids FIRST
- Snacking only (Experimental): Aim: to reduce unhealthy snacking only
  Interventions: Behavioral: Kids FIRST
- Control (No Intervention): Control

INTERVENTIONS:
Behavioral: Kids FIRST — family- and school-based intervention to reduce unhealthy screen-time and snacking
  Arms: Screen-time and Snacking; Screen-time only; Snacking only

SUMMARY:
Kids FIRST was a 12-week, four arm, home- and school-based pilot randomised controlled trial to reduce screen-time and unhealthy snacking with assessments at pre- (baseline) and post-intervention. Four UK schools were randomised to control or one of three interventions - Group 1: targeting reductions in screen-time and unhealthy snacking (ST+Sn), Group 2: targeting reductions in screen-time only (ST), Group 3: targeting reductions in unhealthy snacking only (Sn). Intervention group parents received four online 'sessions' and four packages of resources which were tailored to each intervention group and focused on specific mediators of screen-time and/or unhealthy snacking. Children received four 30-minute lessons during school time, followed by homework activities/challenges. Children and parents reported their own screen-time behaviours, children reported their own snacking behaviours, and completed questionnaires on individual, behavioural, social and physical home environmental variables. Descriptive analyses were undertaken using principles of intention to treat.

DETAILED DESCRIPTION:
The Kids FIRST intervention was performed and reported in accordance with the Consolidated Standards of Reporting Trials extension to randomised pilot and feasibility trials guidelines. The study was approved by the Ethical Advisory Committee of Loughborough University (R15-PO36).

Setting and recruitment Kids FIRST was family based with a school component. The study targeted families with at least one 9-11 year old child. Families were recruited through schools in the East Midlands region of the United Kingdom between September and December 2015. Twenty-five primary schools were selected from a database of schools and school contacts. Headteachers were sent study information via email, which was followed-up with a telephone call, inviting them to be part of the project. In participating schools, parents/caregivers of children aged 9-11 years (year 5 and 6 of Primary School) were sent information sheets via the school outlining the study details and inviting them and their child to participate.

Study design The study was a pilot four-arm cluster randomised controlled trial with assessments at pre- (baseline) and post-intervention (13 weeks after baseline). The study arms were three intervention groups and a control group. The intervention groups were: Group 1: targeting reductions in screen-time and unhealthy snacking (ST+Sn), Group 2: targeting reductions in screen-time (ST), and Group 3: targeting reductions in unhealthy snacking (Sn). Following consent by headteachers, schools were randomised to either one of the three intervention groups or the control group by NP using computer generated random sequences. Only NP had access to the randomisation sequences (which were on a password protected file). This method of randomisation eliminated the possibility of contamination between pupils and parents from the same school.

Theoretical underpinning of the Kids FIRST intervention The Kids FIRST intervention was framed in a social ecological perspective, and was theoretically informed, drawing on constructs designed to address potential individual, behavioural, social and physical home environmental mediators derived from Habit Theory, Behavioural Choice, and Social Cognitive theories of individual behaviour change.

The taxonomy of behaviour change techniques was applied to characterise the association between the potential mediators targeted in the Kids FIRST study, the intervention components / strategies developed, and the theoretical underpinning. Supplementary Table 1 describes the specific behaviours that were targeted by the intervention and the practical application of the behaviour change techniques applied in relation to the Kids FIRST intervention.

Kids FIRST intervention overview The intervention was implemented over a 12-week period from October 2015 to May 2016 (rolling recruitment of schools) following the baseline assessments. Families in each of the three intervention arms received the same structure of intervention, but the content was tailored to the targeted behaviour(s). Parents and children attended an introductory group session at school which provided an overview of the programme. Families in the control group did not receive any resources or engage with any sessions. No changes to the trial methods were implemented after the commencement of the programme.

Family setting The intervention consisted of four blocks of three weeks. Each block targeted and focused on specific evidence-based mediators. All intervention families were given access to the Kids FIRST website (which was live for the duration of the study only), which included a login page where families were directed to the content/pages that were specific to their intervention group (i.e. families in group 1 could only access the webpages for group 1) by a group sensitive password. During each block, parents in each intervention group received one online session, and a package of resources (e.g. newsletters, information sheets, charts etc.) delivered via their child from school. The online sessions introduced the topic of the block to the parents and were followed by the newsletters and resources which prompted 'try at home' activities and challenges with a focus on the specific mediators. Online sessions were delivered via PowerPoint or an audio file and were focused on providing parents with support in the form of informational and cognitive, behavioural, environmental, and social support intervention components as a means of empowering families to make behavioural changes that were specific to them. The newsletters and resources (e.g. monitoring charts, top tips, recipes, and alternative activity or snack ideas) aimed to support the key learning messages delivered in the online sessions and to the children in the classroom lessons (see below).

The key messages of the programme, which were reinforced at each block of the intervention, were:

* Increase knowledge about ST/Sn outcomes (health and other);
* Increase awareness and implementation of strategies to participate in healthy ST and/or consumption of healthy snacks
* Guide parents on how to implement behaviour modification, such as planning and monitoring.

School setting Children randomised to an intervention received four 30-minute lessons during school time over the intervention period (one per 'block'). Key learning messages incorporating key principles of behaviour change were delivered to whole year group classes by trained research personnel. The class lessons were followed by homework activities/challenges and were aimed at the children and were designed to (i) target habits and self-efficacy, (ii) target screen-time and/or nutritional knowledge; (iii) introduce alternative activities/snacks, and (iv) encourage role modelling. Lessons were designed with class teachers prior to the commencement of the programme and incorporated literacy and numeracy aspects that were aligned to the national curriculum specific for each age group.

ELIGIBILITY:
Inclusion Criteria:

The study targeted families with at least one 5-6 and/or 9-11 year old child.

Exclusion Criteria:

-

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Time spent engaged in screen-time | 3 months
  minutes per week engaged in sedentary screen-time
Frequency of consumption of energy-dense snack foods, fruits and vegetables | 3 months
  Daily frequency of consumption of energy-dense snack foods

SECONDARY OUTCOMES:
Time parents spend engaged in screen-time | 3 months
  minutes per day that parents engaged in sedentary screen-time
parent consumption of energy-dense snacks | 3 months
  Daily frequency of consumption of energy-dense snack foods

IPD SHARING:
Plan to Share IPD: Undecided
Unsure

REFERENCES:
- [Derived] Pearson N, Biddle SJH, Griffiths P, Sherar LB, McGeorge S, Haycraft E. Reducing screen-time and unhealthy snacking in 9-11 year old children: the Kids FIRST pilot randomised controlled trial. BMC Public Health. 2020 Jan 29;20(1):122. doi: 10.1186/s12889-020-8232-9. PMID 31996192